CLINICAL TRIAL: NCT02791074
Title: Non-invasive Determination of Intra-left Ventricular Pressure-time Profile for Diagnosis of Heart Failure With Normal and Reduced Ejection Fraction.
Brief Title: Heart Failure Ventricular Pressure Time Profile
Acronym: HF-VFM
Status: Completed | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/365/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — pro-brain natriuretic peptide (1-76)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Healthy Volunteers will undergo the following studying procedures:
  Echocardiography Arterial tonometry
  Interventions: Other: Echocardiography; Other: Arterial tonometry
- Heart Failure Patients: Patients will undergo the following studying procedures:
  NTproBNP Echocardiography Arterial tonometry
  Interventions: Other: NTproBNP; Other: Echocardiography; Other: Arterial tonometry

INTERVENTIONS:
Other: NTproBNP — To assess its level in the blood, as a marker of heart failure presence and severity.
  Groups: Heart Failure Patients
Other: Echocardiography — To measure heart chamber size, heart function, blood vessel size and blood vessel function. These measurements will help us understand the type and severity of heart failure.
Other: Arterial tonometry — A noninvasive method to obtain arterial pressure waveform.

SUMMARY:
This proposed study aim to:

1. Determine intra-LV pressure-time profile non-invasively using recently developed echo Doppler VFM analysis and applanation tonometry and myocardial elastic properties, in HF subjects (both HFNEF and HFREF) compared to normal volunteers.
2. Correlate calculated intra-LV pressure parameters with NT ProBNP levels.

DETAILED DESCRIPTION:
Heart failure (HF) is a common disease and its syndrome is difficult to diagnose. HF with reduced ejection fraction (HFREF) may be diagnosed based on impaired LVEF (<50%). However, diagnosis of HF with normal ejection fraction (HFNEF) is mainly based on the presence of signs and symptoms.

Central to diagnosis of HF is estimation of intra-cardiac pressure, which can only be obtained from invasive catheterization.

This proposed study aim to:

1. Determine intra-LV pressure-time profile non-invasively using recently developed echo Doppler VFM analysis and applanation tonometry and myocardial elastic properties, in HF subjects (both HFNEF and HFREF) compared to normal volunteers.
2. Correlate calculated intra-LV pressure parameters with NT ProBNP levels.

ELIGIBILITY:
Inclusion Criteria:

* Either

  1. has presented to hospital with a primary diagnosis of Heart Failure or
  2. is attending a hospital clinic for management of Heart Failure within 6 months of an episode of decompensated heart failure, which either:

     * resulted in a hospital admission (primary diagnosis) or
     * was treated in out-patient clinic
* LVEF >50% is used as cut-off value for HFNEF and LVEF < 50% for HFREF.
* NT-proBNP within 7 days of admission > 220pg/ml. If there is no result available, NT-proBNP on the same day as echo scan must be > 220pg/ml.

Exclusion Criteria:

* Haemodynamically significant valve disease defined as more than mild degree of valve stenosis, or more than moderate degrees of mitral or aortic valve regurgitation.
* History of valvular disease, i.e. rheumatic heart disease and/or having undergone valvular replacement.
* Isolated right heart failure due to pulmonary disease.
* Presence of haemodynamically significant obstructive lesions of left ventricular outflow tract.
* History of any organ transplant or who was on a transplant list (life expectancy < 6 months at time of enrollment).
* Presence of end-stage renal failure.
* Pregnancy.
* The patient is unable to provide written informed consent.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 35 diagnosed heart failure patient will be recruited from primary care clinic, outpatient clinics and hospital ward from NHCS.
  40 Healthy Volunteer control group.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-05; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Thu Thao Le, PHD, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No